CLINICAL TRIAL: NCT02104219
Title: A Retrospective, Non-interventional, Epidemiologic Study of the Natural History of Patients With Juvenile-onset Hypophosphatasia (HPP)
Brief Title: Retrospective, Non-interventional Natural History of Patients With Juvenile-onset Hypophosphatasia (HPP)
Status: Completed | Type: Observational
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALX-HPP-502; NCT02104206 (obsolete NCT alias)
Record Dates: First submitted 2014-03-25; First posted 2014-04-04 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Hypophosphatasia (HPP)
Keywords: Hypophosphatasia; HPP; bone disease; Soft Bones; low Alkaline Phosphatase; genetic metabolic disorder; alkaline phosphatase; tissue non-specific alkaline phosphatase; rickets; osteomalacia
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases; Rickets; Osteomalacia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize the natural history of HPP in patients with Juvenile-onset HPP.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a life-threatening, genetic, and ultra-rare metabolic disease characterized by defective bone mineralization and impaired phosphate and calcium regulation that can lead to progressive damage to multiple vital organs, including destruction and deformity of bones, profound muscle weakness, seizures, impaired renal function, and respiratory failure. There are no approved disease-modifying treatments for patients with this disease. There is also limited data available on the natural course of this disease over time, particularly in patients with the juvenile-onset form.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent unless patient is deceased
* Patients with Juvenile-onset HPP, defined as documented onset of first signs/symptoms at ≥ 6 months to ˂18 years
* Documented diagnosis of HPP as indicated by skeletal manifestations and low alkaline phosphatase or genotyping

Exclusion Criteria:

* Received treatment with asfotase alfa in the ENB-006-09 study and/or currently enrolled in the ENB-008-10 study
* Received other treatment and/or intervention to treat HPP up to 15 years old
* Other clinically significant disease

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Juvenile-onset HPP (≥ 6 months and ˂18 years)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (9):
  - Atlanta, Georgia
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Springfield, Missouri
  - St Louis, Missouri
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Houston, Texas
  - Seattle, Washington
- Sydney, Australia
- Winnipeg, Manitoba, Canada
- France (3):
  - Le Kremlin-Bicêtre
  - Paris
  - Toulouse
- Rotterdam, Netherlands
- Moscow, Russia
- Istanbul, Turkey (Türkiye)
- United Kingdom (2):
  - Manchester
  - Sheffield

REFERENCES:
- See also: Hypophosphatasia Website — http://www.hypophosphatasia.com
- See also: Hypophosphatasia Website for Health Care Professionals — http://www.hypophosphatasia.com/hcp/
- See also: HPP support group — http://www.magicfoundation.org
- See also: US Hypophosphatasia Group (Soft Bones) — http://www.softbones.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between March 2014 and September 2014. Fifty-four patients were screened and 32 patients were enrolled at 15 centers across the United States, Canada, Australia, Turkey, The Netherlands, and the United Kingdom.
Groups:
- Retrospective Observational: Patients diagnosed with juvenile-onset HPP (ie, documented onset of first signs/symptoms of HPP at ≥ 6 months to < 18 years of age).
Period: Overall Study
Arm/Group | Retrospective Observational
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Diagnosed With Juvenile-onset HPP: Patients diagnosed with juvenile-onset HPP (ie, documented onset of first signs/symptoms of HPP at ≥ 6 months to < 18 years of age).
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Number analyzed (Participants) | 32
Age, Customized [Mean (Standard Deviation); unit: months] — Age at diagnosis
  months | 47 (32.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Australia | 2
  North America | 25
  Europe | 5
Rickets Severity Scale - RSS [Median (Inter-Quartile Range); unit: units on a scale] — The RSS is a 10-point scale, developed for nutritional rickets, that evaluates the degree of metaphyseal cupping and fraying and the proportion of growth plate affected (10 points = severe cupping/fraying, 0 points = absence of cupping/fraying).
  units on a scale | 1.00 [0.00 to 1.50]
Growth Measured by Height Z-score [Median (Inter-Quartile Range); unit: Z-score] — The Z-score indicates the number of standard deviations away from the mean 0. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
  Z-score | -0.86 [-1.57 to -0.62]
Growth Measured by Weight Z-score [Median (Inter-Quartile Range); unit: Z-score] — The Z-score indicates the number of standard deviations away from the mean 0. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
  Z-score | -0.86 [-1.45 to -0.49]

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Global Impression of Change - RGI-C
Description: The RGI-C scale is a 7-point ordinal scale that is used to evaluate musculoskeletal characteristics of HPP (eg, metaphyseal fraying, demineralization of distal metaphyses). The scores range from -3 (severe worsening) to +3 (complete or near-complete healing).
Time Frame: Between Baseline (earliest available, complete, and readable x-ray set) and all available, readable post-Baseline x-ray sets during the period of patients' aged 5 to 15 years, inclusive.
Population: Patients diagnosed with juvenile-onset HPP.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Number analyzed (Participants) | 32
units on a scale | 0.33 [-0.2 to 1.2]
Statistical Analysis 1: Comparison: Patients Diagnosed With Juvenile-onset HPP; Pairs of radiographs were centrally evaluated by 3 independent, blinded pediatric radiologists trained in the assessment of the skeletal manifestations of HPP. The mean RGI-C score across the 3 radiologists was calculated and served as the patient's RGI-C score for a specific time point; Test type: Superiority or Other; p = 0.0755, Sign test — The p-value is based on a nonparametric sign test used to determine whether the median RGI-C score differs from 0 for each time interval. No multiple comparisons or multiplicity adjustments were conducted

2. Secondary Outcome: Change in Height Z-score From Baseline to Last Assessment
Description: Height measurements were assigned to Z-scores which were calculated using the Centers for Disease Control and Prevention (CDC) 2000 growth charts and methodology. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
Time Frame: Any available growth data during the period of patients' aged 5 to 15 years, inclusive. Baseline is the earliest available assessment while post baselines are time points after Baseline during the defined age period.
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Number analyzed (Participants) | 32
Z-score | -0.05 [-0.31 to 0.34]
Statistical Analysis 1: Comparison: Patients Diagnosed With Juvenile-onset HPP; The earliest documented height measurement that was abstracted within the period from 5 to 15 years of age, inclusive, was defined as the baseline height. Height measurements were assigned to Z-scores calculated using Centers for Disease Control and Prevention 2000 growth charts and methodology. Changes in height Z-score from Baseline were computed by subtracting baseline height Z-score from post baseline height Z-scores. The post baseline time points were grouped by time intervals; Test type: Superiority or Other; p = 0.6344, Sign test — The p-value is based on a nonparametric sign test used to determine whether the median change in height Z-score from baseline to last assessment differs from 0. No multiple comparisons or multiplicity adjustments were conducted

3. Secondary Outcome: Change in Weight Z-score From Baseline to Last Assessment
Description: Weight measurements were assigned a Z-score which was calculated using the Centers for Disease Control and Prevention (CDC) 2000 growth charts and methodology. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Higher Z-scores indicate a better outcome.
Time Frame: as for outcome 2
Population: All patients who met all of the inclusion and none of the exclusion criteria were defined as the enrolled population, which was also the analysis population.
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Number analyzed (Participants) | 32
Z-score | 0.12 [-0.31 to 0.60]
Statistical Analysis 1: Comparison: Patients Diagnosed With Juvenile-onset HPP; The earliest documented weight measurement that was abstracted within the period from 5 to 15 years of age, inclusive, was defined as the baseline weight. Weight measurements were assigned to Z-scores calculated using Centers for Disease Control and Prevention 2000 growth charts and methodology. Changes in weight Z-score from Baseline were computed by subtracting baseline weight Z-score from post baseline weight Z-scores. The post baseline time points were grouped by time intervals; Test type: Superiority or Other; p = 0.4520, Sign test — The p-value is based on a nonparametric sign test used to determine whether the median change in weight Z-score from baseline to last assessment differs from 0. No multiple comparisons or multiplicity adjustments were conducted

4. Other Pre Specified Outcome: Rickets Severity Sale - RSS
Description: The RSS is a 10-point scale, developed for nutritional rickets, that evaluates the degree of metaphyseal cupping and fraying and the proportion of growth plate affected (10 points = severe cupping/fraying, 0 points = absence of cupping/fraying).
Time Frame: Any available data during the period of patients' aged 5 to 15 years, inclusive. Baseline is the earliest available assessment value during the period.
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Number analyzed (Participants) | 32
units on a scale | 0.00 [0.00 to 0.50]
Statistical Analysis 1: Comparison: Patients Diagnosed With Juvenile-onset HPP; The Baseline x-ray set defined for RGI-C, which was compared with its subsequent x-ray sets, was also used as the Baseline x-ray set for the RSS reading. Changes from Baseline were computed based on this baseline RSS score, and postbaseline time points were grouped by intervals of time from Baseline; Test type: Superiority or Other; p = 0.4545, Sign test — The p-value is based on a nonparametric sign test used to determine whether change from baseline in the median RSS score differs from 0 for each time interval. No multiple comparisons or multiplicity adjustments were conducted

ADVERSE EVENTS:
Time Frame: No adverse event data were collected during this retrospective noninterventional study.
Arm/Group | Patients Diagnosed With Juvenile-onset HPP
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in a multicenter study involves a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis. Therefore, PIs are subject to certain disclosure and publication limitations.